CLINICAL TRIAL: NCT00855855
Title: Surveillance for Rates of Hib Disease Among Persons 0 Through 59 Months of Age Receiving Pentacel® or Other Hib Vaccines
Brief Title: Surveillance Program to Determine Product Specific Rates of Invasive Hib Disease
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: M5A15
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Haemophilus Infections; Diphtheria; Tetanus; Polio; Pertussis
Keywords: Diphtheria; Tetanus; Pertussis; Poliovirus types 1-3; Haemophilus influenzae type b; Pentacel®
MeSH Terms: conditions — Haemophilus Infections; Diphtheria; Tetanus; Poliomyelitis; Whooping Cough | interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; pentacel; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; COMVAX; Haemophilus influenzae-type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hib vaccine: Participants has received at least one dose of an Hib vaccine
  Interventions: Biological: DTaP-IPV/Hib

INTERVENTIONS:
Biological: DTaP-IPV/Hib — 0.5 mL, Intramuscular
  Other Names: Pentacel®; ActHIB™; Comvax™; PedvaxHIB™

SUMMARY:
To monitor the occurrence of invasive Hib disease over time and to determine product-specific rates of invasive Hib disease within the monitored population.

DETAILED DESCRIPTION:
The purpose of the study is to conduct surveillance for Hib disease.

Prospective active population-based surveillance for invasive Hib disease, conducted by the Center for Disease Control and Prevention (CDC) Active Bacterial Core (ABCs) program within geographic regions currently representing 12% of the US population, will provide Hib case-occurrence (numerator) data.

The ABCs program and the National Center for Health Statistics will provide annual estimates of the number of persons under surveillance, by age group, within the ABCs catchment area.

Ongoing telephone sample surveys, conducted by M/A/R/C, a national sampling organization, will provide brand-specific vaccine exposure data by age group within the ABCs program catchment area at appropriate pre-specified intervals (denominator data).

ELIGIBILITY:
Inclusion Criteria:

* Residence within the geographic scope of Active Bacterial Core surveillance (ABCs) during the period of surveillance
* Aged 0 through 59 months (prior to 5th birthday) on the day of inclusion for Hib disease surveillance and 2 through 23 months (prior to 2nd birthday) for Hib vaccine brand usage survey.
* 2009-2014 calendar years inclusive.
* For the Hib vaccine usage survey, agreement to complete the required survey.

Exclusion Criteria:

Not applicable.

Max Age: 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 5.2 million person years over the 6 year study period
Sampling Method: Non-Probability Sample
Enrollment: 20830 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The rate of invasive Hib disease among persons within the population monitored by the Active Bacterial Core surveillance program. | Up to 6 years post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (59):
- United States (59):
  - Albany, California
  - Martinez, California
  - San Francisco, California
  - Applewood, Colorado
  - Aurora, Colorado
  - Brighton, Colorado
  - Castle Rock, Colorado
  - Denver, Colorado
  - Hartford, Connecticut
  - Adamsville, Georgia
  - Auburn, Georgia
  - Canton, Georgia
  - Carrollton, Georgia
  - Cartersville, Georgia
  - Conyers, Georgia
  - Covington, Georgia
  - Cumming, Georgia
  - Dallas, Georgia
  - Decatur, Georgia
  - Douglasville, Georgia
  - Fayetteville, Georgia
  - Good Hope, Georgia
  - Griffin, Georgia
  - Hampton, Georgia
  - Jasper, Georgia
  - Jonesboro, Georgia
  - Marietta, Georgia
  - Newnan, Georgia
  - Annapolis, Maryland
  - Saint Paul, Minnesota
  - Santa Fe, New Mexico
  - Albany, New York
  - Amsterdam, New York
  - Avon, New York
  - Batavia, New York
  - Bellona, New York
  - Canandaigua, New York
  - Catskill, New York
  - Chatham, New York
  - Geneva, New York
  - Mechanicville, New York
  - Medina, New York
  - Palmyra, New York
  - Rochester, New York
  - Schenectady, New York
  - Schoharie, New York
  - Troy, New York
  - Salem, Oregon
  - Ashland City, Tennessee
  - Charlotte, Tennessee
  - Chattanooga, Tennessee
  - Franklin, Tennessee
  - Gallatin, Tennessee
  - Knoxville, Tennessee
  - Lebanon, Tennessee
  - Memphis, Tennessee
  - Murfreesboro, Tennessee
  - Nashville, Tennessee
  - Springfield, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com